CLINICAL TRIAL: NCT01436786
Title: Guided Imagery Effects on Pregnancy Symptoms and Outcomes
Brief Title: Effectiveness of Guided Imagery Intervention on Factors Associated With Maternal Stress and Preterm Birth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 12900; 5P30NR011403 (NIH)
Record Dates: First submitted 2011-09-06; First posted 2011-09-20 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Preterm Birth; Maternal Stress
Keywords: cytokines; Guided imagery
MeSH Terms: conditions — Premature Birth | interventions — Imagery, Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Guided Imagery Intervention (Experimental): The 12 week intervention consists of a set of 4 GI compact discs (CDs), each 20 minutes in length. Participants will be instructed to listen to the CD once a day in a recommended order for weeks 1-4 and used in any order for weeks 5-12.
  Interventions: Other: Guided Imagery
- Control group (No Intervention): continues usual plan of care

INTERVENTIONS:
Other: Guided Imagery — The 12 week intervention consists of a set of 4 GI compact discs (CDs), each 20 minutes in length. Participants will be instructed to listen to the CD once a day in a recommended order for weeks 1-4 and used in any order for weeks 5-12.
  Arms: Guided Imagery Intervention

SUMMARY:
Demonstrating the effectiveness of an economical and feasible intervention such as guided imagery on factors associated with preterm birth, along with better understanding of pathways leading to adverse birth outcomes has tremendous health, social, and financial benefits. This project has the potential to significantly advance the field of nursing and knowledge development in the areas of maternal stress reduction in African American women and to provide scientific evidence of the effectiveness of guided imagery.

DETAILED DESCRIPTION:
Preterm birth (PTB) is the leading cause of neonatal morbidity and mortality and has tremendous health and economic costs for the infant, family, and society. There has been little success in reducing PTB; rates are at an all time high. Of particular concern is the major racial disparity in PTB rates; African American women have the highest proportion of PTB compared to women of other races or ethnicities. There is growing evidence suggesting that PTB may be the end point of sub-acute or chronic pathophysiological changes that occur before clinical symptoms of preterm labor are present. There is also evidence to suggest that psychosocial factors such as maternal stress and the related symptoms of fatigue, anxiety, depression, as well as unhappiness about the pregnancy are associated with negative birth outcomes. It is proposed that these behavioral factors could influence birth outcomes through two possible pathways: (1) a neuroendocrine pathway in which maternal stress may lead to early and/or greater activation of the maternal-placental-fetal endocrine systems, with CRH playing a key role, thereby promoting labor; and/or (2) immunologic or inflammatory pathways which may promote labor through pro-inflammatory mechanisms. Experts agree primary prevention interventions are needed to address the issue of PTB. Guided imagery (GI) has been effective in decreasing self-reported measures of stress, depression, and fatigue as well as influencing neuroendocrine and immune measures in the general population. However, there are only limited studies examining the effects of GI on maternal stress, neuroendocrine measures, and/or birth outcomes, and there are no published studies examining the effect of GI as a primary prevention intervention to improve birth outcomes by reducing stress and related symptoms and influencing the proposed immunologic pathway to PTB. The specific aims of this randomized clinical trial are (1) to test the effects of a GI intervention on maternal stress (perceived stress), related symptoms (fatigue, anxiety, depression, and unhappiness), neuroendocrine (CRH) and immunological mediators (IL-1β, IL-6, Il-8, IL-10, IL-12, TNF-α, IFN-γ, G-CSF, GM-CSF), and birth outcomes (gestational age and neonatal birthweight) in African American women; and (2) to test the proposed theoretical model by examining predicted relationships among stress, fatigue, anxiety, depression, unhappiness, patterns of neuroendocrine and immunologic factors, and birth outcomes. An analysis of covariance (ANCOVA) model will be used to test for group differences between the GI and control groups. To test the proposed theoretical model descriptive statistics, graphical methods and pairwise correlations will be calculated for all baseline data and canonical correlation analysis will be used to look for relationship among groups of the baseline variables. Demonstrating the effectiveness of an economical, easy to distribute and use, intervention on the psychosocial factors associated with PTB and the proposed pathways leading to adverse birth outcomes has tremendous health, social and financial benefits. This project will provide baseline data for further research to test the biobehavioral efficacy of this intervention in larger samples with multiple races/ethnicities as well as test the model during the postpartum period for maternal well-being and infant development.

ELIGIBILITY:
Inclusion Criteria:

* Being pregnant between 14-17 weeks gestation
* Being African American
* 18 years of age or older
* able to read, write and understand English
* verbalize a source of social support
* self-report of no change in level of stress management strategies used within the last month.

Exclusion Criteria:

* carrying multiples
* have had cervical cerclage
* currently use oral corticosteroids
* have uterine or cervical abnormality
* have dissociative disorders, borderline personalities or psychotic pathology
* have medical and/or pregnancy complications known to impact cytokine levels (e.g., gestational diabetes)
* currently use GI techniques.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2010-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
maternal stress (perceived stress) | baseline
maternal stress (perceived stress) | 8th Week
maternal stress (perceived stress) | 12th Week

SECONDARY OUTCOMES:
neuroendocrine (CRH) and immunological mediators (IL-1β, IL-6, Il-8, IL-10, IL-12, TNF-α, IFN-γ, G-CSF, GM-CSF) | baseline
neuroendocrine (CRH) and immunological mediators (IL-1β, IL-6, Il-8, IL-10, IL-12, TNF-α, IFN-γ, G-CSF, GM-CSF) | 8th Week
neuroendocrine (CRH) and immunological mediators (IL-1β, IL-6, Il-8, IL-10, IL-12, TNF-α, IFN-γ, G-CSF, GM-CSF) | 12th Week

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Jallo, PhD, Principal Investigator — VCU
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States